CLINICAL TRIAL: NCT01860313
Title: Mental Health Training for Elementary Teachers Through Tele-education and Its Impact on the School Atmosphere
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Euripedes C. Miguel, Full Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 573974/2008-0
Record Dates: First submitted 2013-05-07; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Mental Disorders
Keywords: effectiveness; distance learning; mental health
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Web-based interactive educational group (Experimental): This group was submited to the web-based interactive education created for train teachers in child mental health, how to identify mental health problems in children and to know how to deal with problematic children in class.
  Interventions: Behavioral: Web-based interactive education; Behavioral: Text and Video-based education
- Text and Video-based education (Experimental): This group received the material that composed the web-based education environment without any kind of interactivity. This material was composed by some videos about children mental health and a support text.
  Interventions: Behavioral: Web-based interactive education; Behavioral: Text and Video-based education
- Waiting List group (No Intervention): This group was used as control group and did not receive any intervention.

INTERVENTIONS:
Behavioral: Web-based interactive education — An educational program for training teachers and educators to better recognize mental health problems in adolescents and children
  Arms: Text and Video-based education; Web-based interactive educational group
Behavioral: Text and Video-based education — This group received the material that composed the web-based education environment without any kind of interactivity. This material was composed by some videos about children mental health and a support text.
  Arms: Text and Video-based education; Web-based interactive educational group

SUMMARY:
The purpose of this study is to create a web-based interactive educational environment to train elementary teachers, to identify children and adolescents in need of specialized mental health care and give them some advises in managing problematic children in class. After the creation of such an educational environment the psychoeducational project was tested in order to verify it's effectiveness.

DETAILED DESCRIPTION:
Objectives: To develop and test the efficacy of a computer-based training to elementary school teachers of the most common mental health problems.

Outcomes: (a)early identification of the most common mental health problems among children and adolescents, (b)teacher's acquirement of manage skills to better deal with behavior problems and (c)teacher's acquisition of important knowledge to refer students to treatment when necessary.

Method: This research includes two steps: a pilot project (already implemented, whose data will be presented here) and a randomized clinical trial intervention (that will be implemented in a few months).

1. Pilot project, without control group - Comprehended six sessions of educational videos covering basic concepts of mental health stigma and the main disorders that affects children and adolescents followed by discussion forums, quizzes and a conclusion web conferencing with a specialist.
2. A randomized controlled trial with a sample of 176 teachers from nine elementary schools were randomly divided in three groups: a web-based interactive educational group (WBIE), a text and video-based educational group (TWBE) and a waiting list group (WL).

Outcome measures: knowledge, beliefs and attitudes of teachers in mental health and satisfaction with the training received.

Results: The results show that there was an increase in knowledge, attitude changes in mental health and reducing stigma among teachers of web-based interactive educational group. Indeed, comparing the three groups of study participants (WBIE, TVBE and WL), was verified that TVBE group compared with WL group did not show a significant statistical difference (B = 0.957, p = 0.127). Comparing WBIE with WL group, the WBIE answers correctly 1:44 (B = 1.44, p = 0.015). Regarding beliefs and attitudes, WBIE group increased significantly in the ability to identify children with mental health problems, search for mental health information, the ability to recognize colleagues with mental health problems. The average confidence in helping a student with mental health problems also showed increased after psychoeducational intervention in WBIE group.

Discussion: After adjusting educational tools, the methodology and with a bigger sample it's expected to have greater positive results. It's very important to offer teachers a basic apparatus so that they will be able to deal with mental health issues in schools.

ELIGIBILITY:
Inclusion Criteria:

* Primary Public Schools of Campos do Jordão City
* Internet Access

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Knowledge in Child and Adolescents Mental Health, beliefs and attitudes in Child Mental Health | baseline and 1 month (just after the intervention)
  Questions about knowledge, beliefs and attitudes in Child and Adolescents Mental Health applied before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Euripedes Miguel, Full Prof, Principal Investigator — University of Sao Paulo